CLINICAL TRIAL: NCT03425214
Title: Exploration of the Reward System by Functional MRI in Narco-cataplexy Patients With and Without REM Sleep Behavior Disorder
Acronym: NC-TCSP-IRMf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CH MONTLUCON (Unknown); Jacques Lacarin Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-375; 2017-A01974-49 (Other: 2017-A01974-49)
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Narcolepsy; Cataplexy
Keywords: functional MRI; Reward system; REM sleep behaviour disorder; Narco-cataplexy
MeSH Terms: conditions — Narcolepsy; Cataplexy; REM Sleep Behavior Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NC with RBD (Experimental): fMRI and video polysmnography
  Interventions: Other: fMRI; Other: Videopolysomnography
- NC without RBD (Experimental): fMRI and video polysomnography
  Interventions: Other: NC (narcolepsy-cataplexy)
- control group (healthy subjects) (Experimental): fMRI
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — Session will be of about 45 minutes. The reward system will be explore using an experimental task during functional Magnetic Resonance Imaging (fMRI). The name of this task is the"monetary incentive delay task".
  Arms: NC with RBD; control group (healthy subjects)
Other: Videopolysomnography — Video polysomnography will be perform in the sleep center during one night if patient did not have vPSG for 1 year.
  Arms: NC with RBD
Other: NC (narcolepsy-cataplexy) — The investigators hypothesize that NC patients with RBD have a more severe dysfunction of the reward system (hypoactivation of the meso-cortico-limbic pathway) than patients without RBD.
  Arms: NC without RBD

SUMMARY:
Up to 50% of Narcolepsy-cataplexy (NC) patients suffer from REM sleep behavior disorder (RBD), a parasomnia.

A strong link was found between RBD and impulse control disorders (ICD) in Parkinson disease (PD) patients. ICD are thought to be related to a dysfunction of meso-cortico-limbic pathways which belong to the so called ''reward system''.

A recent study in IRMf shows that RBD is associated with impaired reward system.

A strong link was found between these two disorders and therefore we believe that RBD is associated with impaired reward system in NC

The main objective of this study is to evaluate differences in brain activation between NC patients with and without RBD.

The investigators hypothesize that NC patients with RBD have a more severe dysfunction of the reward system (hypoactivation of the meso-cortico-limbic pathway) than patients without RBD.

DETAILED DESCRIPTION:
Type of study: Prospective, case control study.

Number of centers: 3 (Clermont-Ferrand, Vichy and Montlucon)

Patients :

The study will be performed in 66 subjects (22 PD patients with RBD, 22 PD patients without RBD and 22 healthy volunteers, age-and sex-matched without any contraindications to perform an MRI)

Study Performance :

During the first visit (Baseline, inclusion visit, 2 hours), each subject will perform a clinical and neurological examination and neuropsychological assessment (depression by the Beck Depression Inventory (BDI); apathy by the Lille Apathy Rating Scale (LARS), impulsivity by the Urgency, lack of Premeditation, lack of Perseverance, Sensation Seeking scale (UPPS)) Eligible patients will be welcomed for a video Polysomnography in the sleep center, for one night (Month 1, 1 night) and in a subsequent visit at the MRI department for the functional MRI (Month 1, 1 hour). This session will be of about 45 minutes. The reward system will be explore using an experimental task during functional Magnetic Resonance Imaging (fMRI). The name of this task is the"monetary incentive delay task".

ELIGIBILITY:
Inclusion Criteria:

* - Men or women, right handed, 18 to 80 years
* Patients with type 1 Narcolepsy according to the criteria of the International Classification of Sleep, 3rd version, 2014
* Acceptance of the protocol and signature of a written consent
* Social security affiliation

Exclusion Criteria:

* Previous history of psychosis or psychiatric disease
* History of stroke or vascular lesion on MRI.
* Perceptual disorder (vision, hearing) may hinder the realization of the protocols,
* Dementia defined by a score across Montreal Cognitive Assessment (MoCA) <26/30.
* Major depressive state defined by a score scale Beck Depression Inventory (BDI)> 14
* Apathy defined by a score ≥ 14 on the Apathy Scale of Starkstein. Patients with a score ≥ this one will be excluded.
* Usual contraindications to MRI, knowing that no contrast agent injection is performed.
* Pregnant woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure of BOLD signal variation in each region of interest | at Month 1
  BOLD signal variation in each region of interest (ventral tegmental area, accumbens nucleus, limbic cortex, prefrontal cortex) measured during fMRI

SECONDARY OUTCOMES:
reaction time to the task | at Month 1
performance score to the task | at Month 1
Beck Depression Inventory score measured during fMRI | at baseline
Lille Apathy Rating Scale score measured during fMRI | at baseline
impulsivity score by the Urgency measured during fMRI | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Livia FANTINI, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France